CLINICAL TRIAL: NCT01960673
Title: The Influence of Head and Neck Position About Oropharyngeal Leak Pressure and Sealing Between the Laryngeal Mask and Vocal Cord Using Different Types of Supraglottic Airway Device
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201306042RIND
Record Dates: First submitted 2013-09-24; First posted 2013-10-10 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: the Influence of Oropharyngeal Leak Pressure and Sealing Between the Mask and Vocal Cord During Changing Patient's Head and Neck Position
Keywords: supraglottic airway,igel-LMA, ambu-LMA, changing position, head and neck position, oropharyngeal leak pressure,degree of rotation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- LMA proseal (Experimental): The investigator will use proseal LMA in this study. The cuff of the proseal LMA could be inflation. It is thought to fix the larynx shape.
  The investigator wants to test the efficacy during 30,45,60 degree of head and neck position.
  Interventions: Device: LMA proseal
- igel LMA (Experimental): igel LMA did not have cuff. The shape, softness and contours accurately mirror the perilaryngeal anatomy.
  The investigator want to test the efficacy of the igel at 30,45,60 degree of head and neck position.
  Interventions: Device: igel LMA
- air Q LMA (Experimental): The air-Q LMA should be used routinely as a classic passive airway. It is user-friendly, placement in patients is easy and air movement is outstanding. It has the added benefit of allowing for intubation using standard ET Tubes.
  It also has the cuff and the contour of the mask is thought to mimic the the shape of the perilaryngeal region.
  The investigator want to test the efficacy of the air Q LMA at 30,45,60 degree of the head and neck position.
  Interventions: Device: air Q LMA
- ambu LMA (Experimental): ambu LMA is also an cuff device LMA. The investigator wanted to test the efficacy about the leak pressure and the view at 30,45,60 degree of head and neck position.
  Interventions: Device: ambu LMA

INTERVENTIONS:
Device: LMA proseal — It would be used to observe the leak pressure at 30,45,60 degree of the head and neck position and the condition between the vocal cord and peri-laryngeal region. The cuff pressure would be kept at 30 cm H20.
  Arms: LMA proseal
Device: igel LMA — It would be used to observe the leak pressure at 30,45,60 degree of the head and neck position and the condition between the vocal cord and peri-laryngeal region.
  Arms: igel LMA
Device: air Q LMA — It would be used to observe the leak pressure at 30,45,60 degree of the head and neck position and the condition between the vocal cord and peri-laryngeal region. The cuff pressure would be kept at 30 cm H20.
  Arms: air Q LMA
Device: ambu LMA — It would be used to observe the leak pressure at 30,45,60 degree of the head and neck position and the condition between the vocal cord and peri-laryngeal region. The cuff pressure would be kept at 30 cm H20.
  Arms: ambu LMA

SUMMARY:
Generally, the laryngeal mask airway is not considered in the surgery which should be changing position in the perioperative period. The shape of the pharynx changes during the head and neck movement and there is probably also a change in the force transmitted to the cuff along the airway tube. Besides, there is evidence that supraglottic airway device can be displaced with rotation. In this article, the investigators want to discuss about that oropharyngeal leak pressure and sealing between the mask and vocal cord while changing head and neck position in perioperative period using different types of supraglottic airway device.

DETAILED DESCRIPTION:
The investigators select adult patients,who are 20-80yrs old and ASA physical status I or II, receiving minor surgery, ex: breast surgery or cystoscope, participated in this randomized cross-over trial. Patients were excluded if they were in the above condition. The patient is at high risk of aspiration, ex:obesity, pregnancy upper GI bleeding or not enough fasting time. The patient could not open mouth or upper airway obstruction. The patient receive major surgery, ex: heart, brain, lung, liver, kidney surgery. The patient has abnormal heart and lung function.

The patient received different types of supraglottic airway device like proseal LMA,ambu LMA, air Q LMA or igel LMA by draw, then the patients will be divided into different groups.In the preoperative period, the investigators documented oropharyngeal leak pressure in these selected positions: neutral position( 0 degree),and rotation 15, 30,45, 60 degrees, etc. However, oropharyngeal leak pressure was measured by closing the expiratory valve of the circle system at fixed O2 flow 3L/min and 20 cm H2O. If the ambu bag is flattening, the investigators will think the leakage happened between the laryngeal mask and our vocal cord. Then the investigators use fiberscope to observe the condition between the epiglottis and the laryngeal mask.

The investigators wanted to compared the mean leak pressure at different head and neck rotation position,ex:neutral,30,45,60 degrees,by using many different types of supraglottic airway device.

The observers define the relationship between epiglottis and vocal cord to describe the condition when the patient is at different degree of head and neck position. Grade I is vocal cord completely visible. Grade IIA is only partially vocal cord visible and epiglottis noted. Grade IIB is no vocal cord visible and only epiglottis noted. Grade III is other condition, ex:trapped epiglottis or no epiglottis visible.

ELIGIBILITY:
Inclusion criteria:

* 20-80 yrs old and ASA physical status I or II,
* Receiving minor surgery, ex: breast surgery or cystoscope

Exclusion criteria:

* The patient is at high risk of aspiration, ex:obesity, pregnancy upper GI bleeding or not enough fasting time.
* The patient could not open mouth or upper airway obstruction
* The patient receive major surgery, ex: heart, brain, lung, liver, kidney surgery.
* The patient has abnormal heart and lung function.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the leakage happened between the laryngeal mask and our vocal cord | If the ambu bag is flattening during the surgery, the observers check the leak pressure between the laryngeal mask and our vocal cord
  The oropharyngeal leak pressure was measured by closing the expiratory valve of the circle system at fixed O2 flow 3L/min and 20 cm H2O. If the ambu bag is flattening, the observers will think the leakage happened between the laryngeal mask and the vocal cord

SECONDARY OUTCOMES:
Use fiberscope to observe the sealing between the mask and vocal cord while changing head and neck position in perioperative period using different types of supraglottic airway device. | During the surgery
  The observer uses the fiberscope to observe the sealing between the vocal cord and epiglottis.

CONTACTS AND LOCATIONS:
Overall Officials: Cihmin Liu, Principal Investigator — anesthesiology department,National Taiwan University hospital
Locations (1):
- Department of anesthesiology,National Taiwan University Hospital, Taipei, Taiwan